CLINICAL TRIAL: NCT02613169
Title: Preventing Mycobacterium Tuberculosis Infection in HIV-Exposed Infants
Brief Title: Infant TB Infection Prevention Study
Acronym: iTIPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Grace John-Stewart, Professor, Global Health, Medicine, Epidemiology, Pediatrics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000341
Record Dates: First submitted 2015-09-16; First posted 2015-11-24 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-03

CONDITIONS: Tuberculosis
Keywords: M. tuberculosis infection; isoniazid; HIV-exposed infants
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoniazid (Experimental): Isoniazid (INH) ~10 mg/kg (7-15 mg/kg), will be administered once daily to infants in INH arm for 12 months.
  Interventions: Drug: Isoniazid
- No Isoniazid (No Intervention): No INH will be administered to this arm.

INTERVENTIONS:
Drug: Isoniazid — HIV-exposed uninfected infants will be randomized to receive either INH or no INH daily for 12 months for the prevention of Mycobacterium tuberculosis (MTB) infection.
  Other Names: INH
  Arms: Isoniazid

SUMMARY:
Randomized controlled trial (RCT) of isoniazid (INH) vs. no INH to prevent Mycobacterium tuberculosis infection in HIV-exposed uninfected (HEU) infants.

DETAILED DESCRIPTION:
The purpose of this trial is to determine whether isoniazid (INH) reduces the risk of Mycobacterium tuberculosis (MTB) infection in HIV-exposed but uninfected (HEU) children, as well as to determine epidemiologic and immunologic correlates of MTB infection in HEU.

ELIGIBILITY:
Inclusion Criteria:

* HIV exposed infants
* Aged 6 weeks within (+ 4 weeks)
* Born to HIV-infected mothers
* Not premature and over 2.5 kg

Exclusion Criteria:

* Infants with known exposure to active TB in household
* Premature and < 2.5 kg

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2016-08; Primary Completion 2019-10 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace John-Stewart, MD, PhD, Principal Investigator — University of Washington, Dept of Global Health
Locations (1):
- Kisumu County Hospital, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zar HJ, Cotton MF, Strauss S, Karpakis J, Hussey G, Schaaf HS, Rabie H, Lombard CJ. Effect of isoniazid prophylaxis on mortality and incidence of tuberculosis in children with HIV: randomised controlled trial. BMJ. 2007 Jan 20;334(7585):136. doi: 10.1136/bmj.39000.486400.55. Epub 2006 Nov 3. PMID 17085459
- [Background] Madhi SA, Nachman S, Violari A, Kim S, Cotton MF, Bobat R, Jean-Philippe P, McSherry G, Mitchell C; P1041 Study Team. Primary isoniazid prophylaxis against tuberculosis in HIV-exposed children. N Engl J Med. 2011 Jul 7;365(1):21-31. doi: 10.1056/NEJMoa1011214. PMID 21732834
- [Result] LaCourse SM, Escudero JN, Mecha J, Warr AJ, Richardson BA, Carimo N, Cranmer LM, Maleche-Obimbo E, Matemo D, Kinuthia J, Hawn TR, John-Stewart G. Cumulative Mycobacterium tuberculosis Infection Incidence (Measured Primarily by Tuberculin Skin Test) Among Infants With Human Immunodeficiency Virus Exposure: Observational Follow-up of an Isoniazid Prophylaxis Trial. Clin Infect Dis. 2022 Dec 19;75(12):2253-2256. doi: 10.1093/cid/ciac393. PMID 35607710
- [Derived] LaCourse SM, Richardson BA, Kinuthia J, Warr AJ, Maleche-Obimbo E, Matemo D, Cranmer LM, Mecha J, Escudero JN, Hawn TR, John-Stewart G. A Randomized Controlled Trial of Isoniazid to Prevent Mycobacterium tuberculosis Infection in Kenyan Human Immunodeficiency Virus-Exposed Uninfected Infants. Clin Infect Dis. 2021 Jul 15;73(2):e337-e344. doi: 10.1093/cid/ciaa827. PMID 32564076
- [Derived] LaCourse SM, Richardson BA, Kinuthia J, Warr AJ, Maleche-Obimbo E, Matemo D, Cranmer LM, Escudero JN, Hawn TR, John-Stewart GC. Infant TB Infection Prevention Study (iTIPS): a randomised trial protocol evaluating isoniazid to prevent M. tuberculosis infection in HIV-exposed uninfected children. BMJ Open. 2020 Jan 21;10(1):e034308. doi: 10.1136/bmjopen-2019-034308. PMID 31969368

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Isoniazid | No Isoniazid
Started | 150 | 150
Completed | 132 | 133
Not Completed | 18 | 17
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 0 | 5
Not completed — HIV | 0 | 2
Not completed — No TB infection endpoint | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isoniazid | No Isoniazid | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 150 | 150 | 300
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] | 6.3 [6.0 to 6.6] | 6.3 [6.0 to 6.4] | 6.3 [6.0 to 6.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 71 | 142
  Male | 79 | 79 | 158
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kenya | 150 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Mycobacterium Tuberculosis (MTB) Infection
Description: Among HEU infants enrolled at approximately 6 weeks of age, compare the risk of acquiring MTB infection during 1 year of follow-up in infants randomized to receive INH vs. no INH using an interferon-gamma release (IGRA) QuantiFERON-TB Gold Plus (QFT-Plus) assay or tuberculin skin test as part of a composite endpoint to determine MTB infection status
Time Frame: at 12 months post randomization
Population: Final analysis 132 in Isoniazid (14 without endpoint and 4 discontinued) and 133 in No Isoniazid arm (9 without primary endpoint, 8 discontinued)
Measure: Number; unit: participants
Arm/Group | Isoniazid | No Isoniazid
Number analyzed (Participants) | 132 | 133
participants | 10 | 18

2. Secondary Outcome: Severe Adverse Events (SAE)
Description: Number of infants with grade 3 or higher treatment-related adverse events as assessed by DAIDS Table for the Grading Severity of Pediatric Adverse Experiences
Time Frame: Over 12 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Isoniazid | No Isoniazid
Number analyzed (Participants) | 150 | 150
Participants | 21 | 16

3. Secondary Outcome: Combined Outcome of MTB Infection, TB Disease, and Death
Description: Number of infants with a combined endpoint of MTB infection, TB disease, and death
  * MTB infection as measured by IGRA or tuberculin skin test at 12 months post-enrollment
  * TB disease including microbiologically confirmed (culture or Xpert positive), or probable TB (clinical diagnosis).
  * Death of infant
Time Frame: Over 12 months after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Isoniazid | No Isoniazid
Number analyzed (Participants) | 146 | 142
Participants | 11 | 19

4. Secondary Outcome: Combined Outcome of MTB Infection Including IGRA, TST, and Additional Interferon-gamma-independent Immune Markers in QFT-Plus Supernatants
Description: Number of infants with MTB infection as measured by
  * IGRA, or
  * Tuberculin skin test (>10 mm) at 12 months post-enrollment, or
  * Interferon-gamma-independent immune markers in QFT-Plus supernatants
  Combined outcome will be defined as positive if IGRA OR TST OR interferon-gamma-independent marker is positive and combined outcome will be defined as negative if none of these is positive (if children do not have all three markers the definition will hold for available markers).
Time Frame: Over 12 months after randomization
Reporting Status: Not Posted

5. Primary Outcome: Mycobacterium Tuberculosis (MTB) Infection Cumulative Incidence
Description: as for outcome 1
Time Frame: at 12 months post randomization
Measure: Number; unit: TB infections/100 person years
Arm/Group | Isoniazid | No Isoniazid
Number analyzed (Participants) | 132 | 133
TB infections/100 person years | 7.0 | 13.4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study, for two years, two months.
Description: Adverse events include Grade ≥3 severe adverse events by DAIDS scale
Arm/Group | Isoniazid | No Isoniazid
All-Cause Mortality (participants affected / at risk) | 0/150 | 1/150
Serious Adverse Events (participants affected / at risk) | 21/150 | 16/150
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isoniazid (N=150) | No Isoniazid (N=150)
HIV infection (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia/URTI (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Gastroenteritis (Gastrointestinal disorders) | 8 (8) | 3 (3)
Malaria (Infections and infestations) | 12 (12) | 6 (6)
Corrective surgery for spina bifida (Surgical and medical procedures) | 0 (0) | 1 (1)
Corrective surgery for cleft palate (Surgical and medical procedures) | 1 (1) | 0 (0)
Corrective surgery for encephalocele (Surgical and medical procedures) | 1 (1) | 0 (0)
Burns (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT02613169/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT02613169/SAP_001.pdf
  • Informed Consent Form (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT02613169/ICF_002.pdf